CLINICAL TRIAL: NCT00559091
Title: A Phase II Study of Ribavirin in Refractory of Relapsed Acute Myelocytic Leukemia M4 and M5 Subtypes
Brief Title: A Study of Ribavirin to Treat M4 and M5 Acute Myelocytic Leukemia
Acronym: Borden-001
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Principal Investigator, Sarit Assouline, Associate Professor, Department of Oncology, McGill University, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR0620KB; REC:06-112
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Acute Myelocytic Leukemia
Keywords: AML; Acute myelocytic leukemia; leukemia; relapsed; refractory; M4; M5
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia; Recurrence | interventions — Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- I (Experimental): Ribavirin
  Interventions: Drug: ribavirin

INTERVENTIONS:
Drug: ribavirin — Ribavirin will be administered orally, twice daily, in the morning and evening with food. The dose selected is 400 mg AM and 600 mg PM. Intrapatient dose escalations can also be performed in defined circumstances. The maximal dose administered will be 1000 mg AM and 1000 mg PM.
  Other Names: Ribasphere (Three Rivers Pharmaceuticals)

SUMMARY:
The purpose of this study is to determine if ribavirin (a drug commonly used to treat hepatitis C) also has activity in the treatment of patients with refractory or relapsed acute myeloid leukemia (AML) of the M4 and M5 subtype.

DETAILED DESCRIPTION:
The eukaryotic translation initiation factor eIF4E is dysregulated in many human malignancies, including a subset of myeloid leukemia (M4/M5 AML and blast crisis CML). eIF4E overexpression leads to oncogenic transformation. Ribavirin impedes eIF4E mediated transformation in vitro, in primary human specimens and in animal models.

While ribavirin has been used extensively for the treatment of viral hepatitis C and its safety profile has been well defined, it has never been used in patients with AML. This study will establish the efficacy and safety of ribavirin in M4/M5 AML patients. In addition, this study will also include correlative studies to determine the effect of ribavirin on eIF4E activity and eIF4E related pathways in M4/M5 AML patients.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of acute myeloid leukemia (AML), either M4 or M5 subtype de novo or resulting from a transformation from MDS or a myeloproliferative disorder.
* Patients with AML who (a) have failed primary therapy -defined as failing two induction chemotherapies, (b) have relapsed or (c) are not suitable for intensive induction chemotherapy will be eligible. OR
* Patients with AML blast crisis from CML if they are not suitable candidates for intensive induction chemotherapy or have failed imatinib mesylate OR
* Patients with secondary AML after MDS if they are not suitable candidates for intensive induction chemotherapy.
* ECOG 0,1,2, or 3
* Life expectancy > 12 weeks.
* Adequate renal and hepatic function

Exclusion Criteria:

* Uncontrolled central nervous system involvement by AML
* Active cardiovascular disease as defined by NYHA class III-IV categorization.
* Intercurrent illness or medical condition precluding safe administration of ribavirin.
* Received any previous therapy within 28 days prior to study entry.Hydrea is permitted but must be stopped 7 days prior to starting study drug.
* Known infection with HIV.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-04; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Measure: Overall response rate | 6 months

SECONDARY OUTCOMES:
Measure: Safety and tolerability, correlative studies | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sarit Assouline, MD, Principal Investigator — Jewish General Hospital; Kathy Borden, PhD, Study Director — Université de Montréal
Locations (3):
- Canada (3):
  - McMaster Hospital, Hamilton, Ontario
  - Maisonneuve-Rosemont Hospital, Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Background] Topisirovic I, Guzman ML, McConnell MJ, Licht JD, Culjkovic B, Neering SJ, Jordan CT, Borden KL. Aberrant eukaryotic translation initiation factor 4E-dependent mRNA transport impedes hematopoietic differentiation and contributes to leukemogenesis. Mol Cell Biol. 2003 Dec;23(24):8992-9002. doi: 10.1128/MCB.23.24.8992-9002.2003. PMID 14645512
- [Background] De Benedetti A, Harris AL. eIF4E expression in tumors: its possible role in progression of malignancies. Int J Biochem Cell Biol. 1999 Jan;31(1):59-72. doi: 10.1016/s1357-2725(98)00132-0. PMID 10216944
- [Background] Kentsis A, Topisirovic I, Culjkovic B, Shao L, Borden KL. Ribavirin suppresses eIF4E-mediated oncogenic transformation by physical mimicry of the 7-methyl guanosine mRNA cap. Proc Natl Acad Sci U S A. 2004 Dec 28;101(52):18105-10. doi: 10.1073/pnas.0406927102. Epub 2004 Dec 15. PMID 15601771
- [Background] Assouline S, Culjkovic B, Cocolakis E, Rousseau C, Beslu N, Amri A, Caplan S, Leber B, Roy DC, Miller WH Jr, Borden KL. Molecular targeting of the oncogene eIF4E in acute myeloid leukemia (AML): a proof-of-principle clinical trial with ribavirin. Blood. 2009 Jul 9;114(2):257-60. doi: 10.1182/blood-2009-02-205153. Epub 2009 May 11. PMID 19433856
- See also: Click here for more information about the study. — http://www.ribatrial.com